CLINICAL TRIAL: NCT00631878
Title: Phase I/II Randomized, Double Blind, Placebo Controlled, Dose Escalation, Safety and Pharmacokinetics Study in VLBW Neonates, a Human Chimeric Anti-Staphylococcal Monoclonal Antibody for the Prevention of S. Epidermidis Infection
Brief Title: Safety and Pharmacokinetics Study in VLBW Neonates With BSYX-A110
Acronym: N002
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biosynexus Incorporated (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Gerald Fischer, MD, President and CEO, Biosyneuxs Incorporated
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MAB-N002
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Neonatal Staphylococcal Sepsis
Keywords: Staphylococcal; Monoclonal antibodies; Very Low Birth Weight Infants; Prophylaxis
MeSH Terms: interventions — pagibaximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)
- 10 mg/kg (Experimental): 10 mg/kg was given on Days 0, 14
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)
- 30 mg/kg (Experimental): 30 mg/kg was given on Days 0, 14
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)
- 60 mg/kg (Experimental): 60 mg/kg was given on Days 0, 14
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)
- 90 mg/kg (Experimental): 90 mg/kg was given on Days 0, 14
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)

INTERVENTIONS:
Drug: Pagibaximab (formerly BSYX-A110) — Pagibaximab at 10, 30, 60, 90 mg/kg intravenously at Days 0 and 14.
  Other Names: BSYX-A110; HU96-110; Pagibaximab

SUMMARY:
"Phase I/II, Randomized, Double Blind, Placebo Controlled, Dose Escalating, Safety and Pharmacokinetics Study in Very Low Birth Weight Neonates of Four Doses of BSYX-A110 for the Prevention of S. epidermidis Infection." The purpose of this study is to evaluate the safety and pharmacokinetics of escalating doses of BSYX-A110 administered on Study Days 0 and 14.

DETAILED DESCRIPTION:
"Phase I/II, Randomized, Double Blind, Placebo Controlled, Dose Escalating, Safety and Pharmacokinetics Study in Very Low Birth Weight Neonates of Four Doses of BSYX-A110, a Human Chimeric Anti-Staphylococcal Monoclonal Antibody for the Prevention of S. epidermidis Infection" will be the first study of BSYX-A110 in the target population of hospitalized, very low birth weight infants. The purpose of this study is to evaluate the safety and pharmacokinetics of escalating doses of BSYX-A110 administered on Study Days 0 and 14.

This will be a randomized, double blind, placebo controlled, dose escalating study of BSYX-A110 in 48 very low birth weight neonates. The dose levels to be evaluated are 10, 30, 60 and 90 mg/kg. Each dose level will enroll 12 infants who will receive two doses of BSYX-A110 or placebo intravenously at a ratio of 2:1 while hospitalized following birth. Infants will be followed for 8 weeks following the first dose of BSYX-A110 or placebo. The primary objective of this study is to evaluate safety and tolerability. The secondary objective is to analyze the pharmacokinetics of BSYX-A110. Positive cultures obtained during the study period will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria at the time of first infusion (Day 0):

1. 3-7 days of age, inclusive
2. Birth weight of 700-1300 grams
3. Survival expected for at least 1 week after infusion
4. Inpatient in a Neonatal Intensive Care Unit with intravenous access
5. Written informed consent obtained from the parent(s) or guardian

Multiple gestations:

1. Siblings from multiple gestations may be enrolled if they each meet the entry criteria
2. No more than 4 subjects in any birth weight or dose cohort may be siblings

Exclusion Criteria:

Patients may have none of the following at either the first or second dose:

1. Clinically overt systemic infection, as determined by history, physical examination, culture or laboratory data. Neonates with known or suspected HIV infection but without other active systemic infection are not excluded.
2. Life threatening hemodynamic instability
3. Severe congenital anomalies or genetic disorders (especially any predisposing to cardiac decompensation) as determined by history and/or physical examination and including but not limited to:

   i. Trisomy 13 ii. Trisomy 18 iii. Hypoplastic Left Heart Syndrome iv. Omphalocele v. Gastroschesis vi. Holoprosencephaly
4. Known or suspected hepatic or renal insufficiency
5. Persistent seizure disorder
6. Immunodeficiency other than due to prematurity
7. A history of immune globulin administration prior to first study drug infusion
8. Any history, in the infant subject or its mother, of a hypersensitivity or severe vasomotor reaction to immunoglobulin G, or blood products.
9. Any of the following laboratory findings

   1. BUN or creatinine > 1.5 x upper limit of normal for age
   2. AST (SGOT), ALT (SGPT) or total bilirubin > 1.5 x upper limit of normal age
   3. Direct bilirubin of > 2.0 mg/dL
   4. Hemoglobin < 9.0gm/dL
   5. White Blood Count < 2,000 cells/mm3
10. Currently receiving or recently received other investigational agents that could interfere with conduct or results of this study. Each patient receiving other investigational agents will be reviewed by the investigator or his designee with the Sponsor prior to the patient's entry into the study.
11. Expectation that the patient will not be able to be followed for the duration of the study.
12. Mother with serology positive for hepatitis B surface antigen
13. Receipt of Hepatitis B vaccine since birth

Ages: 3 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2001-11; Primary Completion 2003-05 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability. | 0 - 52 days

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics and positive cultures. | 0 - 52 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Weisman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: Biosynexus Incorporated — http://www.biosynexus.com